CLINICAL TRIAL: NCT03191773
Title: A Prospective, Multicenter, Single-Arm Study of Anti-CD19 CAR-T Cell Immunotherapy for Refractory /Relapsed B Cell Malignancies
Brief Title: A Study of Anti-CD19 CAR-T Cell Immunotherapy for Refractory /Relapsed B Cell Malignancies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Shenzhen Institute for Innovation and Translational Medicine (Other); Guangzhou First People's Hospital (Other); First People's Hospital of Foshan (Other); Dongguan People's Hospital (Other Government); The First Affiliated Hospital of Guangdong Pharmaceutical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-HS-32
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Acute Lymphocytic Leukemia; Chronic Lymphocytic Leukemia; Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anti-CD19 CAR transduced T cells (Experimental): Patients will receive a lymphodepleting preconditioning regimen with Fludarabine and Cyclophosphamide followed by anti-CD19 CAR-transduced T cells.
  Interventions: Combination Product: Drugs and anti-CD19 CAR transduced T cells

INTERVENTIONS:
Combination Product: Drugs and anti-CD19 CAR transduced T cells — Drug: Fludarabine On days -4 through -2, Fludarabine 30mg/m2 (IV) will be infused over 30 minutes.
  Drug: Cyclophosphamide On days -4 through -2, Cyclophosphamide 300-500mg/m2 IV will be infused over 60 minutes followed by fludarabine.
  Biological: Anti-CD19-CAR T cells On day 0, cells will be infused intravenously IV over 20 - 30 minutes.

SUMMARY:
Autologous T cells engineered to express an anti-CD19 chimeric antigen receptor (CAR) will be infused back to patients with refractory /relapsed B cell malignancies, including lymphoma and leukemia. The patients will be monitored after infusion of anti-CD19 CAR-transduced T cells for safety,adverse events, persistence of anti-CD19 CAR-transduced T cells and treatment efficacy.

DETAILED DESCRIPTION:
Despite progress has been made to date in the treatment of patients with B cell malignancies, including leukemia and lymphoma, many patients with relapsed or refractory diseases do not respond to the standard treatments. It has been shown that anti-CD19 CAR-transduced T cells may be an effective approach to treat the relapsed or refractory diseases. The procedure involves collecting PBMCs from the patients and modifying the T cells to attack the malignant B cells. In this trial, autologous T cells engineered to express an anti-CD19 chimeric antigen receptor (CAR) containing the signaling domains of CD28 or 4-1BB and CD3-zeta will be infused back to patients with B cell malignancies, including lymphoma and leukemia. The patients will be pretreated with a lymphodepleting preconditioning regimen before the infusion of anti-CD19 CAR T cells, and will be monitored for safety, adverse events, persistence of anti-CD19 CAR-transduced T cells and the treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a CD19+ B cell malignancy，including relapsed or refractory B cell leukemia and/or B cell lymphoma；
2. Patients must have a measurable or evaluable disease at the time of enrollment, which may include any evidence of disease including minimal residual disease detected by flow cytometry, cytogenetics, or polymerase chain reaction (PCR) analysis；
3. Patients with history of allogeneic stem cell transplantation are eligible, providing 6 months had elapsed from SCT, they have no evidence of active graft-versus-host disease (GVHD) and no longer taking immunosuppressive agents during the treatment;
4. Able to understand and sign the Informed Consent Document；
5. There is no obvious dysfunctions in heart , liver, lung, kidney, and performance status with ECOG < 2；
6. Life expectancy：More than 3 months for leukemia and more than 6 months for lymphoma.

Exclusion Criteria:

1. Patients that require urgent therapy due to tumor mass effects such as bowel obstruction or blood vessel compression；
2. Patients that have active hemolytic anemia；
3. Patients who have uncontrollable infectious diseases within 2 weeks before enrollment;
4. Patients with human immunodeficiency virus (HIV) antibody seropositive;
5. Active infection of Hepatitis B virus and / or hepatitis C virus;
6. Patients with any residual intracranial implants；
7. Coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system；
8. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease)；
9. Concurrent opportunistic infections；
10. Concurrent systemic steroid therapy；
11. History of severe immediate hypersensitivity reaction to any of the agents used in this study；
12. Women of child-bearing potential who are pregnant or breastfeeding；
13. Patients with cardiac atrial or cardiac ventricular lymphoma involvement；
14. Other anti-neoplastic investigational agents currently or within 30 days prior to start of the treatment；
15. Psychiatric patients;
16. Previous treatment with any gene therapy products.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-06-30 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | 24 months
  To evaluate the safety and feasibility of the administration of anti-CD19 CAR transduced T cells in patients with refractory /relapsed CD19+ B cell malignancies.
Number of participants with clinical responses | 24 months
  To determine if the treatment regimen can result in clinical regression of B cell malignancies in the patients as described above.

SECONDARY OUTCOMES:
Evaluation of overall survial | 24 months
  To evaluate overall survial(OS) after administration of anti-CD19 CAR transduced T cells in patients with refractory /relapsed CD19+ B cell malignancies.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Feng, MD, Study Director — Second Affiliated Hospital of Guangzhou Medical University; Mingjun Wang, MD, Study Director — Shenzhen Institute for Innovation and Translational Medicine
Locations (5):
- China (5):
  - Department of Hematology, Dongguan People's Hospital, Dongguan, Guangdong
  - Department of Hematology, the First People's Hospital of Foshan, Foshan, Guangdong
  - Department of Hematology, Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Department of Hematology, The First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - Department of Hematology,the Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No